CLINICAL TRIAL: NCT03637621
Title: Distal Humerus Fractures: A Data Analysis on Patients Undergoing Open Reduction and Internal Fixation for the Surgical Management of Distal Humeral Fractures
Brief Title: Retrospective Analysis on Distal Humerus Fractures
Acronym: (DHFx)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Orthopaedic Research & Innovation Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ORIF.003
Record Dates: First submitted 2018-07-24; First posted 2018-08-20 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Distal Humerus Fracture
MeSH Terms: conditions — Humeral Fractures, Distal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ORIF — open reduction internal fixation of the distal humerus

SUMMARY:
The purpose of this study is to evaluate preoperative objective measurements for distal humerus ORIF patients and operative objective measurements to determine if there is any effect to postoperative outcomes. Patients who were 18 years old or greater at the time of surgery were followed clinically and radiographically to determine best practice and optimal treatment and technique, risk and rate of complication, and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. >18 years of age
3. Open reduction internal fixation surgical management of a distal humeral fracture performed by principal investigator at St. Elizabeth Healthcare

Exclusion Criteria:

1. Non-English speaking
2. <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible patients of the names principal investigator receiving open reduction and internal fixation of the distal humerus for any indication at St. Elizabeth Healthcare on or after January 1, 2010 will be evaluated and included in the data analysis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
total operative time | preoperative to up to 8 years postoperative
  minutes
amount of blood loss | preoperative to up to 8 years postoperative
  mls

SECONDARY OUTCOMES:
Patient Outcomes | preoperative to up to 8 years postoperative
  American Shoulder and Elbow Surgeon score to measure shoulder function and pain. Scale of 0-100, 100 being the best possible score
Patient Outcomes | preoperative to up to 8 years postoperative
  Simple Shoulder Test score to measure shoulder function. Scale from 0-12, 12 being the most functional.

CONTACTS AND LOCATIONS:
Overall Officials: R M Greiwe, MD, Principal Investigator — The Orthopaedic Research & Innovation Foundation
Locations (1):
- The Orthopaedic Research & Innovation Foundation, Edgewood, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided